CLINICAL TRIAL: NCT02587364
Title: An Oral, Rising, Multiple-Dose Tolerance, Pharmacokinetic and Pharmacodynamic Study of Gemcabene Capsules in Healthy Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics Study of Gemcabene in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1027-003
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Hypercholesterolemia
Keywords: Pharmacokinetics; Lipid Regulator
MeSH Terms: conditions — Hypercholesterolemia | interventions — gemcabene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Gemcabene 50 mg (Experimental): Gemcabene 50 mg
  Interventions: Drug: Gemcabene 50 mg
- Gemcabene 150 mg (Experimental): Gemcabene 150 mg
  Interventions: Drug: Gemcabene 150 mg
- Gemcabene 450 mg (Experimental): Gemcabene 450 mg
  Interventions: Drug: Gemcabene 450 mg
- Gemcabene 750/600 mg (Experimental): Gemcabene 750/600 mg
  Interventions: Drug: Gemcabene 750/600 mg
- Gemcabene 900 mg (Experimental): Gemcabene 900 mg
  Interventions: Drug: Gemcabene 900 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gemcabene 50 mg — Gemcabene 50 mg once daily (QD)
  Arms: Gemcabene 50 mg
Drug: Gemcabene 150 mg — Gemcabene 150 mg once daily (QD)
  Arms: Gemcabene 150 mg
Drug: Gemcabene 450 mg — Gemcabene 450 mg once daily (QD)
  Arms: Gemcabene 450 mg
Drug: Gemcabene 750/600 mg — Gemcabene 750/600 mg once daily (QD)
  Arms: Gemcabene 750/600 mg
Drug: Gemcabene 900 mg — Gemcabene 900 mg once daily (QD)
  Arms: Gemcabene 900 mg
Drug: Placebo — Placebo once daily (QD)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the multiple-dose pharmacokinetic characteristics and pharmacologic activity of gemcabene.

ELIGIBILITY:
Inclusion Criteria:

* Good health as determined by medical history, physical examination, electrocardiogram (ECG), vital signs, and laboratory assessments
* Body weight: 60-100 kg (desirable)

Exclusion Criteria:

* Use of any medication not considered acceptable by the clinical investigators during the 14-day period before the start of the study (Day 1) ;
* Donation of a unit of blood or participation in a study of investigational or marketed drugs during the 30-day period before the start of the study (Day 1);
* If female, of childbearing potential or lactating;
* History of significant reaction to any fibrate lipid-lowering agent; and
* Significant urine collection of any drug which could interfere with the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 1999-04; Primary Completion 1999-09 (Actual); Study Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 29 days
  Cmax
Pharmacokinetcis | 29 days
  Area Under the Curve (AUC)

SECONDARY OUTCOMES:
Plasma lipid levels - percent change from baseline at Day 29 | 29 days
  percent change from baseline for LDL-C, apolipoprotein B (apoB), total cholesterol (TC), triglyceride (TG), very low density lipoprotein (VLDL-C), high density lipoprotein (HDL-C)
Adverse Events | 29 days
ECG | 29 days
  Clinically Significant Changes
Clinical Laboratory - hematology, chemistry | 29 days
  Clinical Laboratory Abnormalities